CLINICAL TRIAL: NCT02242188
Title: Effect of Iron Supplementation on Psychomotor Development of Non-anemic Exclusively or Predominantly Breastfed Infants: Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Supplementing Iron and Development in Breastfed Infants (SIDBI Study)
Acronym: SIDBI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Anna Chmielewska, MD, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SIDBI study
Record Dates: First submitted 2014-09-14; First posted 2014-09-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Iron Deficiency
Keywords: Breastfeeding; Iron supplementation; Psychomotor development; Safety; infants
MeSH Terms: conditions — Iron Deficiencies; Breast Feeding | interventions — Iron; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron (Experimental): Ferric pyrophosphate (powder preparation in sachets: Actiferol, SunActive Fe, Sequoia, Poland) in a single daily dose. Three doses will be used: 7 mg for infants up to 7 kg of body weight, 10 mg for infants from 7 to 10 kg of body weight, and 15 mg for those exceeding the weight of 10 kg. Caregivers will be instructed to administer the daily dose at the same time of a day, after mixing the content of the sachet with a little amount of breastmilk or milk formula.
  The intervention will last from 4 months to 9 months of age.
  Interventions: Drug: Iron
- Placebo (Placebo Comparator): Maltodextrin prepared in sachets. Caregivers will be instructed to administer the daily dose at the same time of a day, after mixing the content of the sachet with a little amount of breastmilk or milk formula.
  The intervention will last from 4 months to 9 months of age.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Iron — Ferric pyrophosphate (powder preparation in sachets: Actiferol, SunActive Fe, Sequoia, Poland) in a single daily dose. Three doses will be used: 7 mg for infants up to 7 kg of body weight, 10 mg for infants from 7 to 10 kg of body weight, and 15 mg for those exceeding the weight of 10 kg. Caregivers will be instructed to administer the daily dose at the same time of a day, after mixing the content of the sachet with a little amount of breastmilk or milk formula.
  The intervention will last from 4 months to 9 months of age.
  Arms: Iron
Dietary Supplement: Placebo — Maltodextrin (packed in identical sachets as active products)
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
INTRODUCTION Exclusively breastfed infants are at risk of iron deficiency. American Academy of Pediatrics (AAP) recommends iron supplementation in exclusively breastfed infants beginning at 4 months of age. Uncertainty exists regarding the effects of iron supplementation during infancy on neurodevelopmental outcomes in the absence of anemia.

AIM To establish whether psychomotor and mental development is influenced by early iron supplementation in healthy, non-anemic, exclusively or predominantly breastfed infants.

METHODS Healthy term newborns will be recruited shortly after birth. If predominantly breastfed (>50% daily feedings) and non-anemic at 4 months, they will be randomized to receive either an iron supplement (approx.1mg/kg/day) or placebo until 9 months of age. Participants will be assessed with use of Bayley Scales of Infant and Toddler Development (Bayley III) at 12, 24 and 36 months of age.

DETAILED DESCRIPTION:
INTRODUCTION Iron is a nutrient of essential importance to the human organism. It takes part in energy production, oxygen transportation, and DNA synthesis and is indispensable for the development of the central nervous system. Iron is required for the myelination and production of neurotransmitters. It has been well documented that iron deficiency anemia (IDA) impairs child development. If the diagnosis of IDA is delayed, the deficits may be irreversible. Iron deficiency (ID) is the most common single nutrient deficiency and may affect 12% of children < 3 years of age in industrialized countries. ID has the potential to negatively influence psychomotor development. However, a causal relationship is not as clear as for IDA.

Previous studies have suggested that iron supplementation in healthy infants may enhance psychomotor development. A meta-analysis carried out by our group (Szajewska et al. ) aimed to evaluate the effects of iron supplementation in non-anemic pregnant women and in non-anemic healthy children aged <3 years on the mental performance and psychomotor development of children. The authors identified 7 randomized controlled trials (RCTs), 5 of which referred to supplementation during infancy. The polled results of 3 RCTs (n = 561) showed significant improvement on the Psychomotor Development Index (PDI) of the Bayley Scales of Infant Development at approximately 12 months of age in the iron-supplemented group compared with the control group (mean difference: 4.21; 95% CI 2.31 to 6.12). No significant effect of iron supplementation on the Mental Developmental Index (MDI) or behavior was found. Since the meta-analysis was performed, one relevant new study has been published. In this follow-up study, cognitive and school performance was measured at the age of 9 years. In the original study, infants were randomized to receive daily supplementation of iron, zinc, iron and zinc or placebo from 4 to 6 months of age and an assessment of iron and zinc status, as well as growth, was performed. No statistically significant difference in cognitive performance or school performance was reported between the four groups.

Given that ID is a common problem in small children, measures to prevent ID are being taken. According to Committee of Nutrition of the European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN CoN), this should be achieved by the promotion of exclusive breastfeeding, the use of iron-fortified formulas when formula feeding is needed, the postponement of the introduction of whole cow milk as the main drink until the end of the first year of life, and the promotion of consumption of complementary foods rich in iron. More recently, the ESPGHAN CoN concluded that there is no convincing evidence that iron supplements should be provided to normal birth weight, exclusively breastfed infants during the first 6 months of life in populations with a low prevalence of IDA among 6-month-olds. In contrast, the American Academy of Pediatrics (AAP) recommends iron supplementation (1 mg/kg) in exclusively breastfed infants beginning at 4 months of age that should be continued until iron from complementary foods is available. Since in partially breastfed infants iron intake is uncertain, those who receive more than one half of their daily feedings as human milk, should also be supplemented with 1mg/kg iron beginning at 4 months.

Interventional studies of good methodological quality evaluating the role of iron supplementation of infants without anemia on their mental and psychomotor development are still needed.

MATERIALS AND METHODS

This is a randomized, double-blind, placebo-controlled trial.

* Participants Healthy singleton newborns born at term in a university hospital (St. Anna Mazowiecka Hospital, Department of Gynecology and Obstetrics, The Medical University of Warsaw, Poland) will be considered for inclusion. Their mothers will be approached shortly after birth and informed consent will be obtained. Parents will be contacted after approximately 3 months in order to establish weather an infant is being exclusively breastfed. If so, the infant will be randomised to receive either an iron supplement or a placebo from the age of 4 completed months until 9 months of age. Infants will also be recruited in well-baby clinics. Apart from recruitment, all study procedures will be pursued in The Department of Paediatrics, The Medical University of Warsaw, Poland.
* Sample size Sample size was calculated with the main outcome of fine and gross motor scales, cognitive and language development of the Bayley Scales of Infant and Toddler Development (Bayley III). In the previous editions of the test, these elements of the assessment were combined into Psychomotor Developmental Index (PDI) and Mental Developmental Index (MDI). To detect a difference of 5 points between the study groups with a power of 80% and α =0.05, a sample of 91 infants is needed in each study group. To account for 20% of loss to follow up, we aim to recruit 220 infants for the study.
* Interventions Infant in the experimental group will receive ferric pyrophosphate (7mg, 10mg or 15 mg depending on body weight daily, i.e. approx.1 mg/kg/day) or placebo from 4 months to 9 months of age.
* Allocation concealment and blinding A computer-generated randomisation list will be prepared. Blocks of ten will be applied. Randomisation will be stratified by infant's gender. Consecutive randomisation numbers (each number assigned to intervention or placebo in a blinded way) will be given to participants at enrollment. The study products will be delivered to the centre in boxes labelled with the letters A and B (meaning of A and B blinded, information deposited in a sealed envelope in a safe at the administrative part of the department). The boxes will also carry the information on the specific dose (7, 10 or 15mg). Subsequently, the letters A and B will be removed from the boxes by an independent person unrelated to the study planning and conduct, and replaced with numeric codes corresponding to the randomisation numbers, e.g. 001 - 7mg, 001 - 10mg, 001 - 15mg, 002 - 7mg, 002 - 10mg, 002 - 15mg etc. Sachets containing the study product will be packed in small packages of 30 pieces each. Neither the collective packages, nor the sachets will carry any labelling and all the unused sachets will always be returned by parents before switching to higher dose. The active product and placebo will be packed in identical sachets and the content will look and taste the same. Researchers, caregivers, outcome assessors, and a person responsible for the statistical analysis will be blinded to the intervention until a statistical report for the 12-months' developmental assessment is available. After that, both the caregivers and main outcome assessor will remain blinded until the completion of the study. The information on intervention assignment will be stored in a sealed envelope in a safe in the administrative part of the department.

ELIGIBILITY:
Inclusion Criteria:

* Term singleton infants (>37 weeks gestational age)
* Birth weight > 2500g
* Healthy at inclusion
* Breastfed exclusively or predominantly (>50% meals) at inclusion
* No previous iron supplementation
* No previous blood transfusion
* Informed consent given

Exclusion Criteria:

* preterm delivery (<37 weeks of gestation)
* birth weight < 2500 g
* multiple pregnancy
* major illness or congenital anomaly
* being <50% breastfed at the time of inclusion
* food allergy
* anaemia (Hb <105 g/L [10.5 g/dL]) at inclusion, lack of informed consent

Ages: 16 Weeks to 18 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Psychomotor development | 12, 24 and 36 months of age
  Psychomotor development will be assessed with the Bayley Scales of Infant and Toddler Development (Bayley III or BSID III) at 12 and 24 months of age.

SECONDARY OUTCOMES:
Hematological and iron status | 4, 12 and 24 months
  Samples will be analyzed for hemoglobin (Hb) concentration, mean corpuscular volume (MCV), hematocrit (HCT), reticulocytes (RET) concentration, serum ferritin, hepcidin, soluble transferrin receptor and calculated soluble transfferin receptor ratio (sTfR), reticulocyte hemoglobin.
Growth | 4, 6, 9, 12, 24 and 36 months
  Weight, length and head circumference will be recorded at 4, 6, 9, 12, 24 and 36 months.
Behaviour | 36 months
  Behaviour will be assessed with use of child behavioral checklist (CBCL)
Adverse events | untill 9 months of age (during intervention)
  Parents will be asked to fill out a form of possible adverse events of the intervention daily. The symptoms listed in the form will include diarrhoea, vomiting, constipation, discolouration of the stool, fever, and respiratory tract infections. The forms will be collected at each check-up visit during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Chmielewska, MD, PhD, Principal Investigator — The Medical University of Warsaw
Locations (1):
- Department of Pediatrics, The Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
This has not been discussed in the study team.

REFERENCES:
- [Derived] Svensson L, Chmielewski G, Czyzewska E, Domellof M, Konarska Z, Piescik-Lech M, Spath C, Szajewska H, Chmielewska A. Effect of Low-Dose Iron Supplementation on Early Development in Breastfed Infants: A Randomized Clinical Trial. JAMA Pediatr. 2024 Jul 1;178(7):649-656. doi: 10.1001/jamapediatrics.2024.1095. PMID 38739382
- [Derived] Chmielewska A, Chmielewski G, Domellof M, Lewandowski Z, Szajewska H. Effect of iron supplementation on psychomotor development of non-anaemic, exclusively or predominantly breastfed infants: a randomised, controlled trial. BMJ Open. 2015 Nov 24;5(11):e009441. doi: 10.1136/bmjopen-2015-009441. PMID 26603252